CLINICAL TRIAL: NCT04256642
Title: Comparison of the Erector Spinae Plane Block Versus Intrathecal Morphine on Post-Cesarean Delivery Analgesia
Acronym: ESPCS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Thammasat University (Other)
Responsible Party: Principal Investigator, Albert Moore, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-5732
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Active Comparator)
  Interventions: Drug: Intrathecal morphine
- Erector Spinae Plane Block (Experimental)
  Interventions: Procedure: Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — A nerve block that injects local anesthetic in the Erector Spinae Plane
  Arms: Erector Spinae Plane Block
Drug: Intrathecal morphine — Intrathecal morphine at the time of spinal anesthesia
  Arms: Intrathecal morphine

SUMMARY:
This study is a Randomized Control Trial comparing the Erector Spinae Plane Block with intrathecal morphine for post cesarean delivery analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing scheduled Cesarean delivery

Exclusion Criteria:

* Patients with an ASA score greater than 3
* Allergies to study medications
* Contraindications to neuraxial analgesia
* Patients with chronic pain
* Patients unable to communicate in the study language

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
24 hour area under the curve pain scores | First 24 hour
  It will be measured at 3 6 12 18 and 24 hours after the end of the cesarean delivery. This pain will be assessed by asking the patient to go from lying to sitting (or use incentive spirometry) and rated using a linear 10 cm visual analogue scale (VAS). The 24 hour pain VAS area under the curve (AUC) will be calculated using the trapezoid rule.

SECONDARY OUTCOMES:
Measurement of quality of recovery after cesarean delivery | First 24 hours
  At 24 hours the ObsQoR11, a validated instrument to measure the quality of recovery after cesarean delivery, will be administered to the patient
Nausea and vomiting | First 24 hours
  The incidence of nausea and vomiting will be rated on a 10 cm VAS
Analgesic usage | First 24 hours
  The cumulative use of opioids, expressed as morphine equivalents will be recorded at 24 hours.
Pruritus | First 24 hours
  The incidence of pruritus will be rated on a 10 cm VAS
Incidente of persistent surgical pain | Three months
  Patients will be contacted by telephone 3 months after the cesarean to assess the presence of chronic pain. This will be done using a modification of the brief pain inventory

CONTACTS AND LOCATIONS:
Overall Officials: Albert Moore, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No